CLINICAL TRIAL: NCT04508153
Title: A Prospective Randomized Trial Comparing Efficacy of Pelvic Floor Muscle Training With a Digital Therapeutic Device to Standard Exercises for the Treatment of Stress Urinary Incontinence: A Remote Digital Trial
Brief Title: Pelvic Floor Muscle Training With a Digital Therapeutic Device to Standard Exercises for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Renovia, Inc. (Industry)
Collaborators: OBVIO HEALTH USA, Inc. (Unknown); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OBVIO-REN-001
Record Dates: First submitted 2020-08-05; First posted 2020-08-11 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-01

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: A virtual prospective randomized controlled study to evaluate the efficacy of using the leva® PDHS to perform PFMT (leva arm) compared to standard care of a PFM exercise home program (Kegel arm) for the treatment of SUI or SMUI.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized to either the leva® arm or Kegel arm on a 1 to 1 ratio using block randomization. Prior to initiation of the trial, a randomization sequence will be generated by the ObvioHealth system. Participants will be automatically allocated the next available slot in the sequence at the time of their randomization and assigned to the leva® or Kegel group accordingly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Leva PDHS arm (Other): Upon randomization, subjects randomized to the leva® arm will receive the leva® PDHS, and instructions for how to download the smartphone app to facilitate use of the device. They will be instructed to use leva® based on the in-app training provided.
  Within the app, subjects will be instructed to use the leva® device to perform PFMT according to the training program provided through the smartphone app associated with the device. This entails 2 ½ minute training sessions, three times daily, 7 days per week for a total of 8 weeks.
  Interventions: Device: Leva Pelvic Digital Health System
- Kegel arm (Other): Subjects randomized to the Kegel arm will be provided links to view instructions on how to perform PFMT (written instructions per the handout adapted from Voices for PFD, the patient advocacy arm of the American Urogynecologic Society), as well as an audio/visual didactic instructing them to perform Pelvic Floor Muscle Exercises (PFME) three times daily, seven days per week throughout the 8-week study period.
  Interventions: Other: Kegel exercises

INTERVENTIONS:
Device: Leva Pelvic Digital Health System — Pelvic floor muscle training using the pelvic digital health system to treat pelvic floor disorders, specifically stress urinary incontinence.
  Arms: Leva PDHS arm
Other: Kegel exercises — Pelvic floor muscle training (PFMT), commonly referred to as "Kegel" exercises, is a first line conservative treatment for pelvic floor disorders, specifically stress urinary incontinence (SUI) or stress-predominant mixed urinary incontinence (SMUI).
  Arms: Kegel arm

SUMMARY:
A virtual prospective randomized controlled study to evaluate the efficacy of using the leva® Pelvic Digital Health System (PDHS) to perform PFMT compared to a standard home exercise home program for the treatment of SUI/SMUI. The treatment part of the study lasts eight weeks and has two arms. One group will receive routine care consisting of at-home Kegel exercises, and the other will be provided with a leva® device and instructions for use. Subjects in both groups will be assessed at baseline, then at 4 and 8 weeks for change and improvement of their symptoms. They will also be assessed at 6 and12 months after study completion.

DETAILED DESCRIPTION:
This trial is entirely virtual. No office visits, specific locations, or physical examination will be required. Enrollment may occur from any location in the United States

* A virtual prospective randomized controlled study to evaluate the efficacy of using the leva® PDHS to perform PFMT (leva arm) compared to standard care of a PFM exercise home program (Kegel arm) for the treatment of SUI or SMUI.
* Following completion of e-consent and screening, including an initial bladder diary and introductory phone call to review the study requirements, subjects are considered officially enrolled.
* A series of baseline assessments will be administered to all subjects to evaluate symptom severity, frequency and impact.
* Subjects will then be randomized to either the leva® arm or Kegel arm on a 1 to 1 ratio using block randomization. Prior to initiation of the trial, a randomization sequence will be generated by the ObvioHealth system. Participants will be automatically allocated the next available slot in the sequence at the time of their randomization and assigned to the leva® or Kegel group accordingly.
* Prior to beginning the program, subjects in the Kegel arm will receive printed instructions for PFMT with Kegel exercises. Subjects in the leva® arm will be shipped the leva® digital device, along with instructions for use and how to download the corresponding digital app. Day 1 of the study begins the day following receipt of materials.
* Study population: women with SUI or SMUI.
* The study requires no office visits. All participant data will be entered in the subject's smartphone using a custom designed mobile application. Participants will be able to interact with the app throughout the study period and will be presented with surveys and a voiding diary on a specified schedule during an 8-week treatment period. There will also be expected post-intervention follow up surveys at 6- and 12-months
* Using virtual recruiting, a total of up to 350 subjects will be enrolled in the trial.
* Subjects in both arms will have three scheduled phone calls with study staff during the first two weeks of treatment.
* Subjects can speak to the study staff at any time via an in-app chat function, the phone, or videoconference.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Capable of giving informed consent
* Possess a smartphone capable of interacting with the ObvioHealth and Renovia apps
* Self-reported SUI/SMUI symptoms of ≥ three months duration
* Diagnosis SMUI based on Medical, Epidemiologic and Social Aspects of Aging (MESA) stress symptom score (Percent of total possible stress score) greater than MESA urge symptom score (percent of total possible urge score)
* English speaking
* Postmenopausal, post hysterectomy, or willing to use an acceptable method of birth control for the duration of the study
* Able to complete a bladder diary using the ObvioHealth app
* Able to complete electronic surveys and upload data
* Willing to provide contact information and respond to remote contact: phone calls, text messages, email
* Willing to participate in the 8-week study with follow up at 6-and 12-months, refraining from the pursuit of treatment for Stress UI using other modalities (i.e. will not wear a pessary, participate in pelvic floor Physical Therapy or surgery) during the first 8 weeks

Exclusion Criteria:

* Absence of a vagina, per patient report
* Reports seeing or feeling a vaginal bulge or sensation of vaginal bulge
* Diagnosis of any neuromuscular disease that may contribute to UI (i.e., multiple sclerosis, spinal cord injury, Parkinson's Disease, etc.)
* Non-ambulatory, per patient report
* Currently pregnant or <6 months post-partum per patient report
* Currently (or within the last 1 month) breast feeding
* Prior surgery for stress UI
* Previous PFMT: 2 visits within the last 3 months under a supervised therapeutic plan of care
* Currently taking, or has taken within the last 2 months, medication to treat UI
* Prior augmentation cystoplasty or artificial sphincter
* Implanted nerve stimulator for urinary symptoms, active within the past 60 days
* Participation in another clinical study within 30 days of screening
* Impaired cognitive function per patient report and evaluation of medication list
* Contraindication to the use of a vaginal probe
* Unable to understand instructions on the use of the leva® PDHS
* Unable to operate a smartphone app with use of Bluetooth and Wi-Fi connectivity

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Efficacy - Urogenital Distress Inventory (UDI-6) | Baseline, 4 weeks, 8 weeks, 6 months and 12 months
  UDI-6 is a validated questionnaire assessing symptom presence and degree of bother. It will be used to compare the degree of symptom change in the leva arm vs the Kegel arm within and between groups.
Efficacy - Bladder diaries | Baseline and 8 weeks
  Bladder diaries evaluating the average number of stress-incontinence episodes in 3 days will be compared within and between groups

SECONDARY OUTCOMES:
Survey evaluations of incontinence Pelvic Organ Prolapse Distress Inventory (POPDI-6) | Baseline, 4 weeks, 8 weeks, 6 months and 12 months
  POPDI-6 to assess the impact that pelvic floor disorders have on the health related quality of life in women
Patient Reported perception of general health Short Form-20 (SF-20) | Baseline, 4 weeks, 8 weeks, 6 months and 12 months
  SF-20 survey on the participants perception of their general health.
Self-reported adherence | 4 weeks, 8 weeks
  Visual Analog Score for self-reported adherence to the prescribed therapy, 0% = did not adhere to the prescribed treatment regimen/did not perform any Pelvic Floor exercises to 100% = adhered to the prescribed treatment regimen
Correlations between self-reported adherence and device reported adherence in the leva group | 4 weeks, 8 weeks
  Self-reported adherence and Device-reported adherence in the Leva group will be correlated
Incidence of Treatment-Emergent Adverse Events (Safety and tolerability) | Through study completion, an average of 1 year
  Monitored for adverse events and serious adverse events
Feedback on perception of treatment - likelihood of recommending to a friend | 4 weeks, 8 weeks
  Visual Analog Score of likelihood of recommending to a friend Scale from 0-100%. 0%= Will not recommend to a friend to 100%=Will definitely recommend to a friend.
Feedback on perception of treatment - interest in surgical treatment | 4 weeks, 8 weeks
  Visual Analog Score of interest in surgical treatment for urinary incontinence. Scale from 0-100%. 0%= Not interested at all in surgical treatment to 100%=Extremely interested in surgical treatment.
Survey evaluations of incontinence Colorectal-Anal Distress Inventory-8 (CRADI-8) | Baseline, 4 weeks, 8 weeks, 6 months and 12 months
  CRADI-8 to assess the impact that pelvic floor disorders have on the health related quality of life in women
Survey evaluations of incontinence Pelvic Floor Distress Inventory (PFDI-20) | Baseline, 4 weeks, 8 weeks, 6 months and 12 months
  PFDI-20 to assess the impact that pelvic floor disorders have on the health related quality of life in women
Survey evaluations of incontinence Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-IR) | Baseline, 4 weeks, 8 weeks, 6 months and 12 months
  PISQ-IR to assess the impact that pelvic floor disorders have on the health related quality of life in women
Survey evaluations of incontinence Patient Global Impression of Severity (PGI-S) | Baseline, 4 weeks, 8 weeks, 6 months and 12 months
  PGI-S is the participants description of how their urinary tract condition is currently.
Survey evaluations of incontinence Patient Global Impression of Improvement (PGI-I) | 4 weeks, 8 weeks, 6 months and 12 months
  PGI-I is the participants description on how their urinary symptoms are now, compared with how they were before they began the study.
Survey evaluations of incontinence Pelvic Floor Impact Questionnaire (PFIQ) | Baseline, 4 weeks, 8 weeks, 6 months and 12 months
  PFIQ to assess the impact that pelvic floor disorders have on the health related quality of life in women

CONTACTS AND LOCATIONS:
Overall Officials: Holly Richter, MD PhD, Principal Investigator — University of Alabama at Birmingham; Milena Weinstein, MD, Principal Investigator — Massachusetts General Hospital; Gena Dunnivan, MD, Principal Investigator — University of New Mexico; Noelani M Guaderrama, MD, Principal Investigator — Southern California Permanentae
Locations (3):
- United States (3):
  - University of Alabama *** Virtual Trial May be enrolled from any US Location, Birmingham, Alabama
  - Southern California Permanente Medical Group*** Virtual Trial May be enrolled from any US Location, Irvine, California
  - University of New Mexico *** Virtual Trial May be enrolled from any US Location, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weinstein MM, Dunivan GC, Guaderrama NM, Richter HE. Digital Therapeutic Device for Urinary Incontinence: A Longitudinal Analysis at 6 and 12 Months. Obstet Gynecol. 2023 Jan 1;141(1):199-206. doi: 10.1097/AOG.0000000000005036. Epub 2022 Nov 30. PMID 36701620
- [Derived] Weinstein MM, Dunivan G, Guaderrama NM, Richter HE. Digital Therapeutic Device for Urinary Incontinence: A Randomized Controlled Trial. Obstet Gynecol. 2022 Apr 1;139(4):606-615. doi: 10.1097/AOG.0000000000004725. Epub 2022 Mar 10. PMID 35271539
- [Derived] Weinstein MM, Pulliam SJ, Richter HE. Randomized trial comparing efficacy of pelvic floor muscle training with a digital therapeutic motion-based device to standard pelvic floor exercises for treatment of stress urinary incontinence (SUV trial): An all-virtual trial design. Contemp Clin Trials. 2021 Jun;105:106406. doi: 10.1016/j.cct.2021.106406. Epub 2021 Apr 16. PMID 33866003